CLINICAL TRIAL: NCT07012070
Title: Impact of Wearable Activity Linked Kinetic Therapy on the Walking Performance and Vascular Health in Patients With Peripheral Artery Disease: A Randomized Clinical Trial (the WALK-PAD Trial)
Brief Title: Improving Walking Performance in Patients With Peripheral Artery Disease Through Wearable Activity Trackers
Acronym: WALK-PAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, GuangMing Tan, Assistant professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023.548
Record Dates: First submitted 2025-05-27; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Artery Disease
Keywords: wearables; SET; HBET; PAD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: This is a single-centre, open-labelled, parallel-arm, randomized controlled trial. The target population is patients with a diagnosis of symptomatic PAD as defined by the presence of lifestyle limiting claudication and an ankle-brachial-index (ABI) of <0.9. Participants will be randomized at the ratio of 1:1 to receive SET (control), or HBET enhanced with WAM, and an app-based program installed on their mobile device that provides personalized auto- feedback based on their level of activities and lifestyle (treatment). The proposed sample size will be 70 with 35 patients in each arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SET (Active Comparator): Supervised exercise therapy (SET) is The supervised program is conducted at the research institute under the supervision of a qualified healthcare provider. It consists of 12 weeks of intermittent treadmill walking to moderate to severe claudication pain at a speed of ≈2 mph. WAM will be offered to both intervention and control arms, but the mobile apps will only be installed for the subjects randomized to intervention arm. All subjects will receive from their physicians, according to the guidelines, cardiovascular risk management, cholesterol-lowering medication, antiplatelet therapy, the advice to stop smoking, and modification of other atherosclerotic risk factors that were present5. All borrowed devices will be returned at the end of the study.
  Interventions: Behavioral: supervised exercise therapy (SET); Device: Wearable activities monitor (WAM); Behavioral: Mobile application
- eHBET (Experimental): eHBET enhanced with Wearable Activities Monitor (WAM), and an app-based program installed on their mobile device that provides personalized auto-feedback based on their level of activities and lifestyle (treatment). Patients who are already using a smartwatch capable of the steps count and activity monitor before this study are allowed to use their own devices but are encouraged to switch to the FitBit watch for uniformity of data collection. Patients will be encouraged to wear the watch as often as possible during daytime and during sleep. Data gathered will be automatically transmitted wirelessly to a cloud-based platform provided by the manufacturer. The data from the WAM will be extracted and integrated to the mobile apps, accessible only by the research team and the patient. During the randomization visit, patients will be given simple instructions on how to operate the device and how to connect the device to the mobile apps.
  Interventions: Device: Wearable activities monitor (WAM); Behavioral: enhanced HBET; Behavioral: Mobile application

INTERVENTIONS:
Behavioral: supervised exercise therapy (SET) — Supervised exercise therapy (SET) is a structured program of exercise designed for individuals with peripheral artery disease (PAD) and intermittent claudication (IC). It consists of 12 weeks of intermittent treadmill walking to moderate to severe claudication pain at a speed of ≈2 mph and at a grade equal to 40% of the highest workload achieved during the baseline maximal treadmill test, with intermittent period of rest, for at least 3 times per week with a minimum of 30-45 minutes per session
  Arms: SET
Device: Wearable activities monitor (WAM) — The WAM use in this study is the FitBit Inspire 3 Advanced Activity Tracker (FitBit Inc. San Francisco, CA, USA), which is a commercially available tri-axis accelerometer and heart rate monitor capable of continuous monitoring of heart rate using LED sensor, and activities including daily steps count and derived daily activity level, detection of arrythmia and measuring peripheral capillary oxygen saturation. Fitbit devices connect with HOBBIT-PAD platform which was developed specifically for patients with PAD based on user-centred design. It contains patient education information, instruction for exercise, activity record, and embedded messaging function between the patient and the research team about any technical and clinical issue. Important and thorough customizations will be made to tailor this mobile health platform for this study, which includes the addition of patient education materials on PAD and its management, tips on health eating and lifestyle, and tips on exercise.
Behavioral: enhanced HBET — Instructions for HBET are programmed according to the AHA recommendation on the exercise programs for patients with PAD and are automatically generated by the mobile apps. Patients will be prompted to use the exercise function on the mobile apps at least 3 times per week. Once the exercise function is activated, it will extract the steps counts and the walking pace from the WAM during exercise. Patients will be instructed to walk to maximal claudication symptom before stopping, at which point they will press pause on the WAM which will mark the claudication onset time. After the claudication subside, they can resume walking and resume recording on their WAM. Each exercise session will last for 45 minutes excluding rest periods, but the subject can terminate the exercise before the session ends.
  Arms: eHBET
Behavioral: Mobile application — The mobile apps and mobile platform are adopted from the HOBBIT-PAD platform prototype that was developed specifically for patients with PAD based on user-centred design. This platform contains patient education information, instruction for exercise, activity record, and embedded messaging function between the patient and the research team about any technical and clinical issue. The source code for this platform is publicly available. Important customization will be made to tailor this mobile health platform for this study, which includes addition of patient education materials on PAD and its management, tips on health eating and lifestyle, and tips on exercise. These materials are adopted from the patient education materials available on the Hospital Authority and the AHA website. This information will be periodically sent to the subject's mobile device as a push notification to help them better understand their disease and to promote independent self-care and healthy lifestyle.

SUMMARY:
Peripheral Arterial Disease (PAD) of the lower extremities is common and prevalence of PAD is increasing in our aging population. The presence of PAD is associated with increased cardiovascular morbidity and mortality, reduced physical function and quality of life.

Intermittent claudication is the most common symptom of PAD affecting about 30% of the patients. Supervised exercise therapy (SET) is safe and cost-effective therapy when compared with invasive revascularization, and is recommended as the first-line treatment for symptomatic PAD. However, SET is not readily available in the public healthcare system.

Barriers to SET implementation include demands for healthcare resources and the inconvenience of travelling to designated centre for SET. Home-based exercise therapy (HBET) has been proposed as an alternative to SET as they are more accessible and more acceptable to patients, but the benefits of HBET compared to SET have not been consistently demonstrated in studies. Wearable activities monitor (WAM) have been proposed as an adjuvant to enhance the performance of HBET. However, there is no direct comparison of WAM enhanced HBET to SET. Furthermore, WAMs were mainly used for monitoring in HBET in the previous studies and patient feedback was conducted either in-person or over telephones by the researchers, which challenges the true meaning of HBET. In this study, we aim to evaluate the non-inferiority of personalized self-guided HBET enhanced with WAM and auto feedback mobile apps, to SET, in a randomized-controlled trial of patients with symptomatic PAD.

DETAILED DESCRIPTION:
Peripheral Arterial Disease (PAD) of the lower extremities is common and prevalence of PAD is increasing in our aging population. The presence of PAD is associated with increased cardiovascular morbidity and mortality, reduced physical function and quality of life.

Intermittent claudication is the most common symptom of PAD affecting about 30% of the patients. Supervised exercise therapy (SET) is safe and cost-effective therapy when compared with invasive revascularization, and is recommended as the first-line treatment for symptomatic PAD. However, SET is not readily available in the public healthcare system.

Barriers to SET implementation include demands for healthcare resources and the inconvenience of travelling to designated centre for SET. Home-based exercise therapy (HBET) has been proposed as an alternative to SET as they are more accessible and more acceptable to patients, but the benefits of HBET compared to SET have not been consistently demonstrated in studies. Wearable activities monitor (WAM) have been proposed as an adjuvant to enhance the performance of HBET. However, there is no direct comparison of WAM enhanced HBET to SET. Furthermore, WAMs were mainly used for monitoring in HBET in the previous studies and patient feedback was conducted either in-person or over telephones by the researchers, which challenges the true meaning of HBET. In this study, we aim to evaluate the non-inferiority of personalized self-guided HBET enhanced with WAM and auto feedback mobile apps, to SET, in a randomized-controlled trial of patients with symptomatic PAD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are newly diagnosed with symptomatic claudication as defined by the presence of claudication symptoms elicited by the single claudication question
2. Patients who ABI <0.9 are the primary target population

Exclusion Criteria:

1. Patients is inability to ambulate without walking aids or understand the instruction of exercise
2. Patients have history of previous percutaneous or surgical revascularization of lower limb
3. Patients is presence of critical limb ischemia or gangrene
4. Patients has history of major amputation of the lower limb
5. Patients is presence of other co-morbidities which limit walking ability
6. Patients is presence of cardiovascular instability which includes unstable angina or acute coronary syndrome
7. Patients diagnosed active class III/IV heart failure
8. Patients is inability to operate simple electronic devices
9. Patients is inaccessibility of a mobile network service in the place of residence
10. Patients is unwillingness in sharing individual data to study team
11. Patients is life-expectance less than 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute walk test distance | 12 weeks, 26 weeks
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance in meters covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity

SECONDARY OUTCOMES:
compliance to treatment | 12 weeks, 26 weeks
  Compliance to exercise therapy will be measured as the percentage of participation in the SET session in the control arm, and percentage of exercise program activation in the intervention arm.
change in claudication symptoms | 12 weeks, 26 weeks
  claudication symptoms as measured by the Walking Impairment Questionnaire which was The WIQ is a short, validated questionnaire for patients with peripheral arterial disease that is easy to complete. It contains three domains to assess walking impairment: walking distance, walking speed, and stair climbing. For each domain, a sub-score of the Likert items was calculated. The mean of these domains represents the total WIQ score. The Chinese version of the WIQ has been validated by our centre against the claudication symptoms and showed to be a reliable and clinically relevant instrument
change in quality of life | 12 weeks, 26 weeks
  The 36-items short-form (SF-32) health survey score score will be converted to SF-6D index score which is a preference-based measure of health-related quality of life (HRQoL) for its descriptive ability. The SF-6D index score will be used in the subsequent cost-effectiveness analysis.
change in endothelial function | 12 weeks, 26 weeks
  endothelium function will be evaluated using the Flow-mediated dilatation (FMD). The test will be performed in a quiet, temperature-controlled room with the subject lying supine. Subjects are advised to refrain from ingesting caffeine, high-fat foods and vitamin C or use tobacco for at least 6 hours prior to the study. After a qualified image is acquired for analysis, a pressure cuff placed distal to the imaging probe at the forearm will be inflated to 50mmHg above the systolic pressure for 5 minutes. The longitudinal image of the brachial artery is scan continuous for 3 minutes after the deflation of the cuff. The percentage change in peak brachial artery diameter before and after the cuff inflation will be calculated automatically and reported as the FMD of the subject.
change in arterial compliance | 12 weeks, 26 weeks
  arterial compliance as measured by the carotid-femoral pulse-wave velocity which is is a well-validated surrogate measurement of arteria stiffness and is an important prognostic marker for future cardiovascular event39. Several previous studies have shown a reduction in cfPWV after a period of exercise training in non-PAD individuals. The Vicorder (software version 4; Skidmore Medical) which uses the oscillometric technique to acquire the pulse waveform, will be used for cfPWV measurement. Measurements of cfPWV will be obtained by using a 10-cm-wide cuff around the right upper thigh to detect the femoral pulse and a 3-cm cuff around the neck to detect the right carotid pulse. The distance between the suprasternal notch and mid upper thigh cuff is used as the travel distance between the carotid and the femoral cuff. The cfPWV is calculated automatically as cfPWV (m/s)=distance (m)/transit time (s)
change in lower limb perfusion | 12 weeks, 26 weeks
  lower limb perfusion as measured by Exercise ankle-brachial index (ABI) and Transcutaneous oxygen tension (TcPO2) .Exercise ABI will be performed using the Gardener progressive graded treadmill protocol (2mph, 0% grade with 2% increase every 2 minutes) until maximal claudication pain or for a maximum of 5 minutes. Immediately after exercise, the patient is asked to lie in a supine position and ABI test is repeated. The difference between the resting ABI and post exercise ABI reflects lower limb perfusion on exertion.
change in calf muscle strength | 12 weeks, 26 weeks
  The assessment of isometric muscle strength of the lower extremities will be assessed for knee extension, knee flexion, ankle plantarflexion, and ankle dorsiflexion. All tests will assess the muscle strength by the peak force and the rate of force development using a hand- held dynamometer (microFET2, Hoggan Scientific, Salt Lake City UT, USA) which has been shown to have excellent correlation with the criterion-reference dynamometers42. The presence of PAD significantly weakened lower extremity power43. However, the impact of exercise on muscle strength has not been definitively ascertained44
change in blood inflammatory markers | 12 weeks, 26 weeks
  Blood Tests for cardiovascular risk factors including Haemoglobin A1c as measured in percentage of glycated hemoglobin and lipid profile as measured in mmol/l will be sent to local laboratory for processing. Additional blood tests for high-sensitivity C- reactive protein (hs-CRP) as measured in mg/L, and interleukin-6 (IL-6) as measured in pg/ml will be sent to an accredited medical laboratory for processing as these parameters are not available as a routine blood test at the local laboratory.
cost-effectiveness | 12 weeks, 26 weeks
  Cost-effectiveness analysis will be carried out from a health-care payer perspective, and non health-care consequences such as effects on production loss or cost of transportation to the health-care facility will not be considered. The cost for each treatment will be calculated with reference to the gazetted price from the Hospital Authority. The current listed price for SET is HKD 2830, and the cost for eHBET involves only the WAM which is listed at HKD800. The incremental cost-effectiveness ratio (ICER) will be calculated using between group cost difference divided by difference in HRQoL. Following the World Health Organization's guidelines, we defined the willingness-to-pay (WTP) threshold as 1 times the local gross domestic product per capita (which is US $49,146= HKD 384,284 in 2021), and the treatment is considered cost-effective if the ICER of the treatment is lower than the WTP threshold.
change in skin perfusion | 12 weeks, 26 weeks
  TcPO2 measures the local oxygen released from the capillaries through the skin, reflecting the metabolic state of the lower limb. The reproducibility of TcPO2 is much higher than ABI therefore allowing for a detection of a relatively small changes in lower limb perfusion after any therapeutic intervention. TcPO2 will be measured using the Perimed Periflux System 6000 (Perimed Corporation, Stockholm, Sweden) with the patient lying supine in a well-lit and temperature-controlled room. Two electrodes whose membranes are maintained at 45°C are placed on the dorsum of the foot and equilibration will be allowed before taking any measurement.

CONTACTS AND LOCATIONS:
Overall Officials: GuangMing Tan, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong, Hong Kong
  - Prince of Wales Hospital, Hong Kong, Shatin